CLINICAL TRIAL: NCT07255534
Title: Efficacy and Safety of Digital Therapeutics for Improving Shoulder Function After Rotator Cuff Repair: A Prospective, Randomized, Parallel-Group, Evaluator-Blinded Study
Brief Title: Efficacy and Safety of Digital Therapeutics for Improving Shoulder Function After Rotator Cuff Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JiHye Hwang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMC 2025-07-113-002; RS-2024-00401350 (Other Grant/Funding Number: Korea Health Industry Development Institute)
Record Dates: First submitted 2025-09-28; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Rotator Cuff Tear Arthropathy; Repair of a Cuff Tear
Keywords: Rotator Cuff Tear Arthropathy, repair of a cuff tear, digital therapeutics, rehabilitarion
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled, 1:1 allocation, total participants 70
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrevention group (digital therapeutics) (Experimental)
  Interventions: Other: digital therapeutics; Other: usual care
- control group (usual care) (Active Comparator)
  Interventions: Other: usual care

INTERVENTIONS:
Other: digital therapeutics — After rotator cuff repair surgery, the patient performed prescribed rehabilitation exercises delivered through a personal mobile device
  Arms: Intrevention group (digital therapeutics)
Other: usual care — Before discharge and at the first postoperative visit (2 weeks after surgery), patients receive education based on a brochure covering rehabilitation exercises, surgical site care, and criteria for hospital visits in emergency situations. The brochure includes information on the duration of brace use, surgical site hygiene and care, precautions for arm use, and detailed rehabilitation exercise instructions.
  At follow-up visits around 8 and 20 weeks post-surgery, patients receive guidance on improving joint range of motion and muscle strengthening exercises. Physical therapy modalities such as cold and heat application and electrical stimulation are provided. Additional treatments, including corticosteroid injections combined with hyaluronic acid, may be administered based on the healthcare provider's clinical judgment.

SUMMARY:
1. Importance of Rehabilitation After Rotator Cuff Repair Rotator cuff tears are among the most common shoulder conditions in Korea. They can occur naturally with aging or result from trauma or overuse. When conservative treatments like medication or injections fail to relieve pain and restore function, rotator cuff repair surgery is necessary. Postoperative rehabilitation exercises are crucial for recovering shoulder function, reducing pain, and returning to daily activities. Many studies have emphasized the importance of staged rehabilitation and patient education after surgery, showing that active patient participation directly affects recovery. However, some patients rely on unverified internet sources (such as YouTube or online forums) or face limitations such as time, geographical constraints, or cost even when receiving face-to-face therapy.
2. Advantages of Digital Therapeutics Digital therapeutic devices have emerged as a promising solution to these challenges. These smartphone applications deliver exercise and educational content tailored to postoperative rehabilitation, aiming to improve the disease state. They offer anytime, anywhere access without time or location restrictions and provide evidence-based, systematic, and personalized rehabilitation programs. Comprehensive educational materials enhance patient understanding and promote self-management skills, potentially increasing rehabilitation adherence.
3. Recent Research Findings Digital rehabilitation programs for patients after rotator cuff repair have demonstrated effectiveness. Programs that provide real-time exercise feedback using mobile apps and sensors have shown similar or superior outcomes compared to traditional physical therapy. Augmented reality (AR)-based rehab systems are more effective in improving shoulder function than conventional methods, and digital apps offering customized exercise videos significantly enhance physical function and confidence. Notably, patients using digital rehabilitation programs for 1 to 6 months exhibited improved adherence to therapeutic exercises, facilitating consistent home-based rehabilitation.
4. Purpose of This Clinical Trial While previous studies have confirmed the efficacy and safety of digital therapeutic devices after rotator cuff surgery, most are limited to generic exercise programs. This clinical trial aims to evaluate the effectiveness and safety of a clinical trial digital therapeutic device not yet approved domestically, providing disease-specific exercise programs.

ELIGIBILITY:
Inclusion Criteria:

1. Be an adult aged 19 or older.
2. Have a diagnosis corresponding to Korean Standard Classification of Diseases codes M75.1 (rotator cuff tear) or S46.08 (other specified injuries of tendons and muscles at shoulder and upper arm), and have undergone rotator cuff repair (RCR) surgery, or RCR combined with procedures such as acromioplasty, biceps tenotomy, fixation, or labrum repair.
3. Own a smartphone operating on the Android or iOS platform.
4. Have received a full explanation of this clinical trial, understood it, voluntarily agreed to participate, and provided written consent to comply with study precautions.

Exclusion Criteria:

1. History of previous rotator cuff repair surgery on the same site (revision surgery).
2. Planning or recommendation by medical staff for contralateral rotator cuff repair surgery within one year after enrollment.
3. Plans to receive direct manual therapy or invasive procedures (e.g., oriental medicine treatments, injections, regenerative therapies) at the surgical site through inpatient or outpatient care at another hospital within one year post-discharge.
4. Presence of severe underlying conditions, neuromusculoskeletal disorders, visual impairment, uncontrolled diabetes, cardiovascular disorders, or other comorbidities that hinder participation in rehabilitation exercises.
5. Difficulty using clinical trial medical devices due to cognitive impairment (e.g., dementia), visual impairment, or digital illiteracy.
6. Other cases where the medical staff judges that unsupervised rehabilitation exercise is contraindicated or the principal investigator deems the subject unsuitable for the clinical trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons score (ASES) | baseline, 9-week, 15-week, 22-week, 46-week
  domain : pain, function
  1. Pain is measured using a Visual Analog Scale (VAS) rated out of 10 points and then converted to a 50-point scale.
  2. Function is assessed through a questionnaire consisting of 10 items, each scored from 0 to 3, with a total raw score of 30. This total is converted to a 50-point scale.
  This results in a final combined score ranging from 0 to 100, with higher scores indicating better shoulder function.

SECONDARY OUTCOMES:
Constant score | baseline, 9-week, 22-week, 46-week
  The scoring system ranges from 0 to 100 points, with higher scores indicating better shoulder function. It includes the following components: pain (15 points), activities of daily living (20 points), active range of motion (ROM) (40 points), and muscle strength (25 points). Muscle strength is measured by assessing force in 90-degree shoulder abduction and then converted into a score.
Korean shoulder Score (KSS) | baseline, 9-week, 22-week, 46-week
  The scale ranges from 0 to 100 points, with higher scores indicating better function. It is composed of the following components: pain (30 points), function (40 points), activities of daily living (10 points), muscle strength (20 points), and satisfaction (10 points).
Simple shoulder Test (SST) | baseline, 9-week, 22-week, 46-week
  The score ranges from 0 to 12 points, with higher scores indicating better function. It is an outcome measure consisting of 12 yes/no questions related to function. Each "yes" response is scored as 1 point, and the total number of "yes" answers is summed to calculate the final score. This tool provides a simple patient-reported outcome to briefly assess the ability to perform daily activities.
Shoulder pain (PVAS) | baseline, 9-week, 15-week, 22-week, 46-week
  Evaluated during rest and activity. Pain is assessed using an 11-point scale (0-10 points) evaluating overall shoulder pain over the past 7 days. A lower score indicates an improvement in pain.
Shoulder joint range of motion (active) | 9-week, 15-week, 22-week, 46-week
  A. Forward flexion (0-180 degrees), abduction (0-180 degrees), and external rotation at the side with the upper arm beside the torso (0-90 degrees) are measured using a goniometer to record the maximum angles. Higher values indicate better shoulder mobility.
  B. Internal rotation at the back: When the arm is placed behind the back, the level of the spine reached by the tip of the thumb is measured and scored accordingly (thoracic vertebrae T1-T12 = 1-12 points; lumbar vertebrae L1-L5 = 13-17 points; buttock = 18 points). Higher scores indicate better shoulder mobility.
Shoulder joint range of motion (passive) | baseline, 9-week, 15-week, 22-week, 46-week
  A. Forward flexion (0-180 degrees), abduction (0-180 degrees), and external rotation at the side with the upper arm beside the torso (0-90 degrees) are measured using a goniometer to record the maximum angles. Higher values indicate better shoulder mobility.
  B. Internal rotation at the back: When the arm is placed behind the back, the level of the spine reached by the tip of the thumb is measured and scored accordingly (thoracic vertebrae T1-T12 = 1-12 points; lumbar vertebrae L1-L5 = 13-17 points; buttock = 18 points). Higher scores indicate better shoulder mobility.
Shoulder muscle strength (Isokinetic) | baseline, 22-week, 46-week
  Isokinetic muscle strength is measured for each movement following a standardized protocol using an isokinetic dynamometer (HUMAN NORM; exercise testing and evaluation device; classification number A30130.01, Class 2 medical device). During the test, the subject sits on a chair with the trunk fixed to the dynamometer. The subject holds the handle on the opposite side of the dynamometer. Higher values indicate better muscle strength.
  Internal and external rotation: The arm is abducted to 45 degrees in the scapular plane with the elbow flexed to 90 degrees. External rotation range of motion is set at 65 degrees and internal rotation at 25 degrees. Measurements are taken at an angular velocity of 60 degrees per second for 4 repetitions (strength) and 180 degrees per second for 10 repetitions (muscular endurance), recording peak torque in pounds.
Shoulder muscle strength (Isometric) | baseline, 9-week, 22-week, 46-week
  Using a hand-held dynamometer (FGN-20B, SHIMPO, JAPAN), the maximum force (in pounds) is collected and measured in the internal rotation (at side), external rotation (at side), and scaption positions.
Global change rating (GRoC) | 22-week, 46-week
  The overall change assessment scale ranges from -5 (much worse) to 5 (much improved) points, evaluating the patient's perception of overall functional recovery and satisfaction with their general condition. Compared to pre-surgery, a change of 2 points or more at the end of intervention (T3), and similarly from T3 to the end of follow-up (T4), is interpreted as the minimum clinically important difference.

OTHER OUTCOMES:
Self-efficacy for exercise (SEE) | baseline, 9-week, 15-week, 22-week, 46-week
  The scale consists of 9 items describing situations that hinder exercise. It uses a 0% (not confident at all) to 100% (extremely confident) scale, with intervals of 10%, assessing the patient's confidence in being able to exercise for 20 minutes, three times a week in each situation. Scores are interpreted as follows: 0-20% = not confident at all, 20-40% = slightly confident, 40-60% = moderately confident, 60-80% = very confident, and 80-100% = extremely confident.
World Health Organization Disability Assessment Schedule (WHODAS 2.0) | baseline, 9-week, 15-week, 22-week, 46-week
  The assessment evaluates difficulties experienced over the past 30 days and consists of 36 items covering six core domains: cognition, mobility, self-care, interpersonal relationships, activities of daily living, and social participation. Each item is rated on a 5-point Likert scale from "no difficulty at all (0 points)" to "extreme difficulty or impossible (4 points)." The total score is calculated by summing all domain scores, ranging from 0 to 100 points. Higher scores indicate greater functional difficulty and a higher level of disability, while lower scores represent better function and lower disability.
(K-eHEALS) | baseline
  Health literacy is assessed by measuring the ability to search for, understand, evaluate, and utilize health information. Scores range from a minimum of 8 to a maximum of 40 points, with higher scores indicating better literacy. A score of 24 or below (criteria may vary by study) suggests a high likelihood of difficulty in searching for and using health information on the internet.
System Usability Scale (SUS) | 22-week
  It consists of 10 items designed to evaluate the usability of the system, with a score range from 0 to 100. Higher scores indicate that the system is easier and more convenient to use.
Satisfaction with the clinical trial medical device (mobile application) | 22-week
  A survey is conducted to assess overall mobile app satisfaction, perceived usefulness, perceived ease of use (PEOU), attitude toward using technology, and behavioral intention to use.
  A Likert scale (1-5 points) is used, with higher scores interpreted as indicating a greater likelihood of technology acceptance.
Resource Utilization | 22-week, 46-week
  This investigates the occurrence and frequency of any additional external treatments the patient received aside from the intervention provided by the institution (including visits to other hospitals, imaging tests, physical therapy, injections/procedures, medications, etc.) and collects perceived benefit scores (0-10 points).
  This monitoring helps identify protocol violations and evaluates additional medical and economic burdens between the two groups, potentially revealing cost advantages.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, Republic of Korea, South Korea

IPD SHARING:
Plan to Share IPD: No
Since this provides the subject's personal information to a third party, separate consent is required.